CLINICAL TRIAL: NCT05854108
Title: Comparison of Cervical Traction Versus Snag to Improve Pain and Quality of Life in Cervical Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/535
Record Dates: First submitted 2023-03-18; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Quality of Life; Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Traction (Other)
  Interventions: Diagnostic Test: Cervical Traction
- Snag Therapy (Experimental)
  Interventions: Diagnostic Test: Snag

INTERVENTIONS:
Diagnostic Test: Cervical Traction — Cervical Traction to Improve Pain and Quality of Life in Cervical Radiculopathy
  Arms: Cervical Traction
Diagnostic Test: Snag — Snag to Improve Pain and Quality of Life in Cervical Radiculopathy
  Arms: Snag Therapy

SUMMARY:
For the wellness by Comparing of Cervical Traction Versus Snag to reduce Pain and improve Quality of Life in Cervical Radiculopathy

ELIGIBILITY:
Inclusion Criteria:

* Males and females were included. Age group 20-50 years. Patient suffering with neck pain radiating down the arms. Patients with positive Spurling test, cervical distraction and upper limb tension test.

Exclusion Criteria:

* Subject suffering with any systemic diseases of MSK. Patients already suffering with pain in shoulder and upper extremity which is of local origin.

Patient with cardiovascular or respiratory disease. Patients having osteophytes in cervical vertebrae. Hypermobility of cervical region.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 6 Months
Quality of Life Scale QOL | 6 Months
  QOL to improve Quality of Life in Cervical Radiculopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No